CLINICAL TRIAL: NCT02656628
Title: A Multi-Center Prospective, Observational Patient Registry of the Dynamic Locking Screws in Metaphyseal and Diaphyseal Shaft Fractures of the Humerus, Femur and Tibia
Brief Title: Observational Patient Registry of the Dynamic Locking Screws
Acronym: DLS
Status: Withdrawn | Type: Observational
Why Stopped: Due to the voluntary recall of the study device (DLS 3.7mm and DLS 5.0mm)
Sponsor: Synthes GmbH (Industry)
Collaborators: Synthes Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: STU-TRA-T-08-198-03
Record Dates: First submitted 2014-07-04; First posted 2016-01-15 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Proximal or Diaphyseal Humerus Fracture; Diaphyseal or Distal Femur Fracture; Diaphyseal, Distal or Proximal Tibia Fracture
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fractures of humerus femur tibia: Dynamic Locking Screw 3.7mm and 5.0mm
  Interventions: Device: Dynamic Locking Screw 3.7mm and 5.0mm

INTERVENTIONS:
Device: Dynamic Locking Screw 3.7mm and 5.0mm — Treatment with DLS and locked plate constructs (small or large fragments)

SUMMARY:
The purpose of this multi-center patient registry is to obtain first clinical results and to assess short and mid-term clinical outcome data of patients treated with DLS.

DETAILED DESCRIPTION:
This is a multicenter, open-label non-comparative, observational patient registry conducted at 15 to 20 clinical sites.

Patients who have agreed participate and have signed an informed patient consent prior to surgery will be included. Follow-up visits will be performed at the following time points: baseline (pre-and postoperative), at 6 weeks, 12 weeks, 6 months, and (12) months (for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit).

To minimize potential bias of the observational study design, a reasonable sample of investigators and sites (15-20 sites), and patients (up to 200 patients) are selected. Furthermore, data will be analyzed by an independent Contract Research Organization, and objective outcome measures are used eg, WOMAC, QuickDASH, fracture healing.

All data collected on the electronic case report forms (eCRF) for this registry will be de-identified. Each patient will be assigned to a unique reference number. eCRFs are confidential documents and will only be available to the Sponsor (including Sponsor delegates, like clinical research associates (CRAs), the Investigator, the investigation statistician, and if requested to the advisory committee, ethical committees and regulatory authorities. The key to link the unique reference number to the patient will be kept in the investigation file by the Principal Investigator for each investigation site.

Registry procedures:

Baseline visit/Pre-Op:

* Potential study patients are informed about the study by the Investigator (or delegate)
* All inclusion and exclusion criteria are checked to determine if the patient can participate in the registry
* Prior to any registry-specific examination, the patient gives written informed consent (IC) and the IC form is placed into the patient's medical record. A copy of the IC and the written patient information is handed over to the patient
* Collection of demographic data, medical history (Charlson Comorbidity Score(49;50)), concomitant medications, fracture characteristics and accident/injury information
* Collection of X-rays: all imaging procedures are organized and prepared for the transmission to the Clinical Research Organization (CRO) as outlined in the imaging manual
* Documentation of study-specific questionnaires (QuickDASH, WOMAC, EQ-5D) based on the reported pre-injury status
* The data are entered into the eCRF

Intra- and postoperative procedures:

All surgical procedures will be done per the standard of care at the treating institution. Aftercare and rehabilitation procedures will be left to the surgeons' discretion.

Follow-up visits:

* Post-operative: before hospital discharge
* 6 weeks (7 - 56 days)
* 12 weeks (57 - 120 days)
* 6 month (121 -270 days)
* (12 month (271 - 425)): for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit

The following procedures are performed during these visits:

* Assessment of fracture healing
* Assessment of physical function and symptoms (QuickDASH*, WOMAC*, weight bearing or load on the affected extremity status)
* Screening for AE or serious AE including documentation and reporting
* Documentation and reporting of secondary surgical interventions due to device or procedure related Adverse events
* Assessment of health-related quality of life (EQ-5D*)
* Collection of X-rays
* Data entry into the eCRF.
* Appointment for the next visit

Clinical Investigation Administration:

The clinical investigator(s) will permit registry-related monitoring, audits, ethics committee review and regulatory inspection(s), thereby providing direct access to the facilities, personnel and to source data/documents on request. The Sponsor's staff or representatives will closely monitor the conduct of the registry so that any questions and problems that may arise can be promptly resolved. Such monitoring will also ensure that the registry is conducted in accordance with this registry protocol, including all amendments and with the requirements of national regulations and ISO 14155.

Monitoring will involve periodic visits, by the Sponsor's representative to the investigation site to verify compliance with all requirements of the registry, to observe procedures and to audit the registry for quality control purposes (presence of required documents, informed consent and for comparison of the case report forms with source data). The frequency of these periodic visits will depend on the enrolment rate and whether there are any difficulties in running the registry in a given site. A monitoring plan describes all monitoring procedures in detail.

On-site audits may take place and are independent of and separate from routine monitoring or quality control functions. They may take place at various stages during the registry. The clinical investigator/s will be informed in writing and/or by telephone in a timely manner that an independent audit is to take place along with the scope of the audit, a date and timelines involved. Whenever possible, the auditor will be accompanied by the responsible CRA or Sponsor's representative. The auditor may stay at the registry site as long as deemed necessary.

In order to ensure quality of the data, all relevant registry documents (registry protocol, case report forms, patient information) will be reviewed by a person not involved in the set-up and management of the registry. The results of the audit will be documented in an audit report and any corrective actions needed from the Investigator communicated to the Principal Investigator.

In general, data collected in the hospital patient charts are considered as source data. In order to facilitate data collection at the investigation sites, a set of source worksheets (SW) based on all variables outlined in the registry protocol will be provided. Data that is not routinely documented in the hospital chart is collected on these worksheets and therefore, the worksheet is considered to be the source document and has to be kept at the investigation site accordingly. Data collected on patient and surgeon questionnaires are also considered as source data.

Source data will be entered by site staff into a web-based Electronic Data Capture (EDC) system and managed according to a detailed pre-specified Data Management Plan. The Investigator or site coordinator shall complete the eCRF in a timely manner after a patient's visit ie, not later than 10 days after the occurrence of a documentable event.

Completed eCRFs will be verified against source data (ie, source data verification).

Investigators shall provide access to the hospital files and any other medical source document containing patient's clinical/medical information, to the company representative to allow source document verification.

The clinical Investigator is asked to keep a list with full names of all patients participating in the registry, giving reference to the patient records.

After the completion of the registry, an electronic copy of the data collected at each investigation clinic will be provided.

Radiographic images will be collected as per standard imaging procedures (standard of care) at the investigation site following patient examinations at discharge, 6 and 12 weeks, 6 and (12) months. Digital de-identified images will be sent to GCTM. Transfer of imaging data to GCTM and handling of the de-identified imaging data at GCTM will be performed according to GCTM standard procedures. More details are described in the imaging manual.

Images relevant for the registry will be retained de-identified electronically as part of the TMF in accordance with relevant guidelines.

The central registry database will be monitored by GCTM representative and queries will be made on a regular basis to each participating site as needed to ensure the quality and integrity of the data.

Data management will be performed by GCTM. Data handling and protection are conducted according to the guidelines of International Organization for Standardization (ISO) 14155 and applicable regulations.

A study specific Data Management Plan describes all details of data management and quality control of the study database at GCTM.

All trial-related essential documents (i.e. documents which individually and collectively permit evaluation of the conduct of an observational study and the quality of the data produced) will be retained by the clinical Investigator for at least 15 years after the end of the registry or as per national requirements. In case where this is not possible, the Sponsor will organize archiving facilities for the source data, in accordance with data confidentiality regulations. The Sponsor will inform the clinical investigator(s) in writing when these documents no longer need to be retained.

The Sponsor will retain specific essential documents in the Trial Master File (TMF) according to the relevant guidelines.

The Principal Investigator at each investigation site has the primary responsibility for patients' treatment, follow-up and overall compliance with the registry protocol, national regulatory requirements and the requirements of ISO 14155. It is advisable that the investigation site appoints a study coordinator who can become the primary point of contact for the CRA concerning overall registry administrative matters.

All Investigators using the DLS in the registry must be trained on the registry device, the registry protocol requirements, national regulations and requirements of the ISO 14155 prior to becoming involved in the patient registry and include their curriculum vitae (CV) in the Investigator file with a copy for the Sponsor' TMF. This training shall be documented by the CRA and/or the Principal Investigator on the site personnel log along with the authorized tasks the Principal Investigator delegates to each team member and an identification of signature.

The registry obligations for the Sponsor, the Clinical Research Associate, and the Investigator are followed as outlined in the ISO14155 and any applicable regulation, and reviewed with the Investigator prior to the start of the registry.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Any of the following fracture types:

  * Proximal or diaphyseal humerus fracture
  * Diaphyseal or distal femur fracture
  * Diaphyseal, distal or proximal tibia fracture
* Eligible for treatment with Synthes DLS and locked plate constructs (small or large fragments)
* Patients able and willing to sign informed consent form
* Patients able and willing to adhere to 12-months follow-up visits

Exclusion Criteria:

* Polytrauma
* Pregnant or nursing females
* Patients already participating in an investigational trial
* Patients who are not expected to survive the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the in- and exclusion criteria and have signed an informed patient consent prior to surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic callus formation and location of callus evaluation: Change over time | 6 weeks, 12 weeks, 6 months, and (12)* months
  The radiologic presence of callus at the four locations around the plate is overall evaluated by a central independent trauma fellow or radiologist:
  * Lateral (under the plate)
  * Medial (on the contra lateral cortex)
  * Anterior
  * Posterior
  "*"for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit

SECONDARY OUTCOMES:
Fracture union | 6 weeks, 12 weeks, 6 months, and (12)* months
  The proportion of patients with a healed fracture will be assessed at each follow-up visit. Each investigator will assess locally bone healing according to the following definitions:
  Union is radiographically defined as continuous mineralized bridging callus between the most distal and the most proximal fragments across the fracture site, where fracture lines are obscured.
  Delayed union is defined as insufficient signs of bridging callus ie, healing has not advanced at the average rate for the location and type of fracture.
  Non-union is defined as insufficient signs of bridging callus ie, healing has not advanced at the average rate for the location and type of fracture (>9 months).
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
QuickDASH for patients with humerus fracture | Time point: 6 and 12 weeks, 6 and (12)* months
  The QuickDASH is a shortened version of the disabilities of the arm, shoulder and hand (DASH) outcome measure. Instead of 30 items, it uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The items ask about the degree of difficulty in performing different physical activities because of arm, shoulder or hand problems, the severity of each of the symptoms of pain, tingling, as well as the problem's impact on sleep. Each item has five response options. The score ranges from 0 (no disability) to 100 (most severe disability).
  The pre-injury QuickDASH score will be assessed by asking the patient before surgery to recall the status before the injury. Additionally, the QuickDASH will be completed and compared at each follow-up visit.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
WOMAC for patients with femur and tibia fractures | Time point: 6 and 12 weeks, 6 and (12)* months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a multidimensional self-administered health status instrument to assess the dimensions of pain (five items), joint stiffness (two items), and disability (17 items).
  It is among the most widely used, valid, reliable, and disease specific health outcome measure for the knee function and arthritis. The questions can either be scored on a 5-point Likert scale, on a 100mm Visual Analogue Scale (VAS), or on a 11-box Numerical Rating Scale (NRS).
  In this study, the items will be scored on a 100mm VAS. The WOMAC score ranges from 0 to 96 points, where 0 equals no disability, and 96 equal's maximal disability.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
Full weight bearing or full use of the upper extremity | 6 and 12 weeks, 6 and (12)* months
  The duration of postoperative non-weight bearing or postoperative inability to full use of the upper extremity will be summarized.
  At each follow-up visit the proportion of patients with full weight bearing or full use of the upper extremity without restrictions will be estimated.
  Full weight bearing is defined as the ability to bear the whole body weight on the affected leg.
  Full use of the upper extremity is defined as the ability to use the upper extremity without any restrictions on loading.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
Adverse Events related to the device or procedure | intra-and postoperative; 6 and 12 weeks; 6 and (12)* months
  The proportion of patients who experience adverse events (AE) related to the device or procedure within 6 and (12)* months after surgery will be estimated. The occurrence of any AE related to the device or procedure will be assessed and documented by the Investigator during 6 and (12)* months after surgery.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
General adverse events not related to the device or procedure | postoperative; 6 and 12 weeks; 6 and (12)* months
  The proportion of patients who experience general AEs (not related to the device or procedure) within 6 and (12)* months after surgery will be evaluated. All general AEs will be assessed and documented by the Investigator during 6 and (12)* months after surgery.
  All patients experiencing general AEs must be followed up until the symptoms subside and any clinically relevant changes have returned to baseline, or until there is a satisfactory explanation for the changes observed.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
Secondary surgical interventions due to device or procedure related Adverse events | postoperative; 6 and 12 weeks; 6 and (12)* months
  All secondary surgical interventions will be documented by the Investigator during 6 and (12)* months after surgery.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit
Health related quality of life: EuroQoL (EQ-5D) | Baseline; 6 and 12 weeks; 6 and (12)* months
  The EQ-5D is a standardized instrument for use as a measure of health outcome. It was designed for self-completion covering the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a three-point categorical response scale: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking in the box against the most appropriate statement in each of the five dimensions. Furthermore, health state is indicated by drawing a line from the box to whichever point on the scale indicates how good or bad health state is today. The endpoints on the scale (VAS) are labeled "worst imaginable health state" and "best imaginable health state" anchored at 0 and 100 respectively.
  *for patients with insufficient signs of healing at the 6 months visit; otherwise preferable visit

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Alexandra Hospital, Woolloongabba, Brisbane, Queensland, Australia